CLINICAL TRIAL: NCT02751853
Title: Effects of Acutely Elevated Afterload oN Left VentRicular Contractility and RElaxation in Heart Failure With Preserved and Reduced Ejection Fraction
Brief Title: Effects of Acutely Elevated Afterload on Left Ventricular Contractility and Relaxation
Acronym: ANREP-EF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the heterogeneity in the first group.
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Holger Thiele, Director, Department of Cardiology, Angiology, and Intensive Care Medicine, University Heart Center Luebeck, University of Luebeck
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-011
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HFPEF (Experimental): Patient with heart failure with preserved ejection fraction (HFPEF)
  Interventions: Device: Conductance catheter
- HFREF (Experimental): Patient with heart failure with reduced ejection fraction (HFREF)
  Interventions: Device: Conductance catheter
- No HFPEF/HFREF (Active Comparator): Patient without heart failure with preserved ejection fraction (HFPEF) or heart failure with reduced ejection fraction (HFREF)
  Interventions: Device: Conductance catheter

INTERVENTIONS:
Device: Conductance catheter — Continuous online measurements of left ventricular pressure and volume using conductance catheters

SUMMARY:
Aim of the study is to assess the effects of abruptly increased afterload on left ventricular contractility and relaxation in patients with heart failure with preserved ejection fraction (HFPEF), patients with heart failure with reduced ejection fraction (HFREF), and patients without HFPEF or HFREF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for left and right heart catheterization
* HFPEF (Group 1) OR HFREF (Group 2) OR absent echocardiographic evidence of HFREF OR HFPEF(Group 3)

AND

* Sinus rhythm during invasive measurements
* Age ≥18 years
* Negative pregnancy test in women with childbearing potential
* Written informed consent

Exclusion Criteria:

* Acute coronary syndrome
* Acute myocardial infarction <6 months
* Planned cardiac surgery or cardiovascular intervention within 6 months following inclusion
* Valvular heart disease >2°
* Severe comorbidities with limited life expectancy <12 months
* Precapillary pulmonary hypertension
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Hemodynamic parameter 1: Changes in contractility assessed by the end-systolic pressure-volume relationship | Day 1
  Changes in contractility after handgrip exercise assessed by the end-systolic pressure-volume relationship

SECONDARY OUTCOMES:
Hemodynamic parameter 2: Changes in contractility assessed by the peak power index | Day 1
  Changes in contractility after handgrip exercise assessed by the peak power index
Hemodynamic parameter 3: Changes in relaxation assessed by the relaxation constant "tau" | Day 1
  Changes in relaxation after handgrip exercise assessed by the relaxation constant "tau"
Functional parameter: Changes in ejection fraction | Day 1
  Changes in ejection fraction after handgrip exercise assessed by echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided